CLINICAL TRIAL: NCT06306534
Title: Intraoperative Acute Study to Evaluate Auditory Intranerve Stimulation
Brief Title: Auditory Intranerve Stimulation Study
Acronym: AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AIS-001; CIV-22-05-039592 (Other Grant/Funding Number: Blackrock Neurotech)
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-02

CONDITIONS: Auditory; Nerve
MeSH Terms: conditions — Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insert Array Into Auditory Nerve (Experimental)
  Interventions: Other: Auditory Nerve Acute (ANA) Electrode Array

INTERVENTIONS:
Other: Auditory Nerve Acute (ANA) Electrode Array — To measure eABRs when stimulating the human auditory nerve

SUMMARY:
This feasibility clinical investigation is designed to answer the question of whether auditory brainstem responses can be safely elicited by acute electrical stimulation within the human auditory nerve.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patients who will undergo an acoustic neuroma removal surgery and are functional deaf
3. Age ≥ 18 years
4. Women with childbearing potential: willingness to use a reliable contraceptive method (e.g. copper intrauterine devices or hormonal methods) after consulting their gyncecologists

Exclusion Criteria:

1. Disabilities in addition to hearing impairment which might interfere with the study procedure
2. Pregnant and breast feeding woman or other vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Elicit a typical eABR Wave V with at least 0.2 µV in amplitude and a latency of the peak around 5 ms | 4 weeks

SECONDARY OUTCOMES:
Collection of adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lenarz, Prof. Prof. Dr., Principal Investigator — Hannover Medical School, Director of otorhinolaryngology
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No